CLINICAL TRIAL: NCT03623360
Title: Prediction of Outcomes in Cirrhosis Using Novel Magnetic Resonance Imaging Biomarkers of Liver Function
Brief Title: Functional MRI to Determine Severity of Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Leeds (Other)
Collaborators: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Ian Rowe, University of Leeds Academic Fellow and Honorary Consultant Hepatologist, University of Leeds
Other Study IDs: IRAS 224109
Record Dates: First submitted 2018-08-01; First posted 2018-08-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Liver Cirrhosis; Liver Fibrosis
Keywords: Gadoxetate disodium
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with liver cirrhosis: The cohort includes patients who encompass the full clinical spectrum of liver function within cirrhosis.
  The participants will undergo a full MRI protocol for liver screening including morphological imaging, fibrosis scoring tests based on relaxometry and diffusion maps, and our novel functional technique based on free breathing DCE-MRI.
  Interventions: Diagnostic Test: Free breathing DCE-MRI

INTERVENTIONS:
Diagnostic Test: Free breathing DCE-MRI — Free breathing DCE-MRI

SUMMARY:
This is a pilot study to investigate the feasibility of a novel MRI technique to assess the severity of liver cirrhosis and predict complications based on functionality and perfusion measurements whilst maintaining image quality.

The principal objective of this pilot study is to assess liver function and the future risk of complications in patients with cirrhosis, using novel techniques and measures based on free-breathing Dynamic Contrast Enhanced MRI.

Specifically the investigators will assess:

1. Whether sufficient data can be generated in patients with cirrhosis whilst maintaining image quality, and
2. The dynamic range of DCE-MRI measures in patients with cirrhosis.

This pilot study will, if successful, provide sufficient data to support applications for larger studies to evaluate the clinical utility of a DCE-MRI imaging biomarker in patients with cirrhosis.

DETAILED DESCRIPTION:
This is a pilot study to investigate the feasibility of a novel MRI technique to assess the severity of liver cirrhosis and predict complications based on functionality and perfusion measurements whilst maintaining image quality.

Recruitment:

Twenty (20) patients with cirrhosis who attend the Leeds Liver Unit at St James's University Hospital will be purposively selected by members of the research team who are also part of the usual care team for these patients in advance of scheduled clinic visits. The selection will be in a way to encompass the full clinical spectrum of liver function within cirrhosis.

Scan:

An intravenous cannula will be inserted to the patient's arm by the radiographer, for the automated administration of contrast agent during the scan. The participant will be asked to remain still on his/her back throughout the duration of the scan.

Patients will undergo a full MRI protocol including morphological imaging, fibrosis scoring tests based on relaxometry and diffusion maps, and the novel functional technique.

After the scan:

The participant will not have to attend any extra clinics or scan appointments. The research team (that includes members of the participants ongoing care team) will continue to track the health condition of the participant over a long-term period (5 years) to collect information with regards to clinical events such as hospital admissions, change in treatment, further procedures and death. The clinical follow-up information will be collected as part of routine care through scheduled ongoing outpatient appointments.

The data acquired during the scans will be analysed using a novel method to quantify liver function and the liver images will be reviewed by an expert radiologist to ensure that the quality of these is sufficient for future clinical application. A cross-sectional data analysis will be performed to identify associations between the functional biomarkers and clinical indices for the assessment of liver fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed with liver cirrhosis using standard methods (liver biochemistry, ultrasound based elastography and liver biopsy).

Exclusion Criteria:

* Pregnancy
* Allergy/intolerance to Gadolinium based contrast agents
* Severe renal impairment
* Severe respiratory disease
* Inability to undergone MRI due to the presence of metal or electronic implants affected by the magnetic field.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cirrhosis who attend the Leeds Liver Unit at St James's University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Image quality | Up to 7 days
  The image quality evaluated visually by an expert radiologist using a scoring system. The score levels for the image quality assessments is: 1: non-diagnostic, 2: poor, 3: adequate, 4: good, and 5: excellent.
The dynamic range of the Total Blood Flow biomarker. | Up to 7 days
  Calculation of the dynamic range of the Total Blood Flow biomarker (ml/100ml/min).
The dynamic range of the Arterial Blood Flow Fraction biomarker. | Up to 7 days
  Calculation of the dynamic range of the Arterial Blood Flow Fraction biomarker (%)
The dynamic range of the Extracellular Volume biomarker. | Up to 7 days
  Calculation of the dynamic range of the Extracellular Volume biomarker (ml/100ml)
The dynamic range of the Intracellular Uptake Rate biomarker. | Up to 7 days
  Calculation of the dynamic range of the Intracellular Uptake Rate biomarker (/100/min)
The dynamic range of the Biliary Excretion Rate biomarker. | Up to 7 days
  Calculation of the dynamic range of the Biliary Excretion Rate biomarker (/100/min)

SECONDARY OUTCOMES:
Correlation of DCE-MRI measures with clinical outcomes | Up to 7 days
  The secondary outcome measure is the correlation between our biomarkers and the clinical scores for the prediction of mortality (Child-Pugh score and the Model to End Stage Liver Disease (MELD)).

CONTACTS AND LOCATIONS:
Overall Officials: Ian Rowe, Dr, Principal Investigator — University of Leeds
Locations (1):
- St. James's University Hospital, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
The information about the health and care of the participants may be provided to researchers running other research studies in this organisation and in other organisations. The information will only be used by organisations and researchers to conduct research in accordance with the United Kingdom Policy Framework for Health and Social Care Research. This information will not identify the individuals and will not be combined with other information in a way that could identify the participants.
  The images obtained from the MRI scan may also be shared anonymously with Siemens, Inc - the company who have developed the techniques to allow scans to be done without breath holding. These images may be used to improve the way that the scans are processed as well as in illustrations of the quality of the images that can be obtained using this technique.